CLINICAL TRIAL: NCT03729466
Title: Investigation of the Effects of Clinical Pilates Exercises on Primary Caregivers of Special Needs Children: Randomized Comparative Study
Brief Title: Investigation of the Effects of Clinical Pilates Exercises on Primary Caregivers of Special Needs Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Yazgı Şentürk, Principal Investigator Yazgı Şentürk, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETK00-2018-0154
Record Dates: First submitted 2018-10-30; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Sedentary Lifestyle
Keywords: clinical pilates
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: clinical pilates and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): There will be no intervention for 8 weeks
- Intervention group (Experimental): clinical pilates will be given to the intervention group for 8 weeks
  Interventions: Other: clinical pilates

INTERVENTIONS:
Other: clinical pilates — The intervention group will be performed in clinical pilates 45 to 60 minutes twice a week for 8 weeks.
  Arms: Intervention group

SUMMARY:
The aim of this research is to investigate the effectiveness of clinical Pilates exercises applied to primary caregivers of children with special needs, flexibility, muscle strength, endurance, cardiovascular endurance, fatigue, coping attitudes and quality of life, depression and anxiety.

DETAILED DESCRIPTION:
Individuals participating in the study will be randomly divided into two groups through the randomized allocation software program. The first group will be given Clinical Pilates exercise training, while the second group will be considered as the control group. The exercises will be applied to the group attending the Clinical Pilates exercise training for 45-60 minutes, twice a week for a total of 8 weeks. Each movement will consist of one set and 10 repetitions. In the Clinical Pilates program, equipment and exercises will be gradually increased. Equipment to be used throughout the Clinical Pilates program; Pilates cushion, Elastic resistant band (red, green, blue), Exercise ball (65 cm) In the Clinical Pilates group, the training session will start with the warm-up program, core stabilization training, clinical Pilates exercises will be applied to increase the postural smoothness and strength, and the exercise session will be terminated with the cooling period. The clinical Pilates group will be given 5 key elements of clinical Pilates (Respiratory-Centre focus- Chest placement - Shoulder placement - Head-neck placement) will be explained. No exercise program will be applied to the control group for 8 weeks. A sufficient number of trials will be conducted to enable participants to adapt to the evaluation and treatment. The evaluations will be done as pre-test and post-test for both groups and then the groups will be compared. Individuals who have agreed to participate in the study and have signed the information consent form will be included.

ELIGIBILITY:
Inclusion Criteria:

* Caring for children over 3 years of age≥1 with special needs,
* Caring for the child for at least 6 months, with or without blood connection (mother, father, nan, aunt, sibling, carer, etc.)
* Being between the ages of 18-55,
* Has not had regular exercise in the last 6 months (3 days a week, more than 20 minutes)

Exclusion Criteria:

* Have serious orthopaedic, neurological, rheumatologic and psychiatric problems that may prevent clinical Pilates exercises.
* Pregnancy
* Has had a traumatic injury or surgery in the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2018-10-25 (Estimated); Study Completion 2018-12-05 (Estimated)

PRIMARY OUTCOMES:
Fatigue severity scale | up to 8 weeks
  The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Berkiye Kırmızıgil, Study Director — Eastern mediterrean university
Locations (1):
- Eastern Mediterrean Universty, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Senturk Y, Kirmizigil B, Tuzun EH. Effects of clinical Pilates on the fitness in people with children with disabilities: a randomized controlled trial. J Comp Eff Res. 2021 Apr;10(5):409-422. doi: 10.2217/cer-2020-0108. Epub 2021 Mar 12. PMID 33709771